CLINICAL TRIAL: NCT04900324
Title: Intramuscular Injections of Botulinum Toxin in Lateral Pterygoid Muscle in the Treatment of Temporomandibular Dysfunctions: Studying the Interest of MRI Guidance and Ultrasound Guidance
Acronym: MAUSBOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/554
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mandibular Dysfunction
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI guidance (Experimental): Injections of botulinum toxin performed using MRI guidance
  Interventions: Device: MRI guidance
- Ultrasound guidance (Experimental): Injections of botulinum toxin performed using ultrasound guidance
  Interventions: Device: Ultrasound guidance

INTERVENTIONS:
Device: MRI guidance — Injections of botulinum toxin performed using MRI guidance
  Arms: MRI guidance
Device: Ultrasound guidance — Injections of botulinum toxin performed using ultrasound guidance
  Arms: Ultrasound guidance

SUMMARY:
The main hypothesis is that a significant pain improve (measured with Visual Analogic Scale [VAS]) can be observed after injection of botulinum toxin A, meaning the success of the guidance device.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from muscular TemporoMandibular Dysfunctions (TMD) with clinical diagnosis: myofascial pain, limited opening of the mouth, articular noise.
* >= 18 years old
* with signed informed consent form

Exclusion Criteria:

* articular TMD: arthritis or other inflammatory disease of temporomandibular joint, arthrosis, bone deformation, previous fracture of condylar area ;
* electromyographic hypoactivity, pure muscular diseases ;
* oro-mandibular dystonia ;
* botulinum toxin allergy,
* risk of bleeding
* recent or active infection
* intercurrent antibiotic treatment (drug interaction) ;
* vaccination during the 15 days preceding the injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Pain improvement | Month 2
  Significant improvement of the pain measured with VAS (0 to 10), corresponding to at least 30% decrease of the pain after injection of botulinum toxin A

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MEYER, Md PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHu de Besançon, Besançon, France